CLINICAL TRIAL: NCT04103359
Title: Fatigue in Myelodysplasic Patients : Why Blood Transfusion Does Not Systematically Improve Symptoms? (FITME Study)
Brief Title: Comparison of Lower-risk MDS Patients With and Without Improvements in Fatigue Following Blood Transfusion Therapy
Acronym: FITME
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: inclusion rate too low
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Jean Monnet University (Other); Institut de Cancérologie de la Loire (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2019-0701; 2019-A01877-50 (Other: ANSM)
Record Dates: First submitted 2019-09-24; First posted 2019-09-25 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Myelodysplatic Syndromes
Keywords: Myelodysplatic syndromes; elderly; fatigue; blood transfusion; physiopathology
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MDS patients (Experimental): MDS patients receiving blood transfusion
  Interventions: Other: Physiological tests to measure fatigue level

INTERVENTIONS:
Other: Physiological tests to measure fatigue level — Physiological tests to measure fatigue level

SUMMARY:
At present, it is unclear why some myelodysplastic patients (MDS) receiving blood transfusion therapy exhibit an increase in Hemoglobin (Hb) without a concurrent improvement in fatigue. Research is thus required to elucidate on why fatigue persists in some MDS patients in order to devise strategies to alleviate fatigue in "non-responders" to blood transfusion.

DETAILED DESCRIPTION:
One hypothesis is that patients who exhibited persistent fatigue following a blood- transfusion- induced increase in Hb have an impaired ability to utilize oxygen at the peripheral level. This could be the consequence of impairments in vascular function, mediated by endothelial dysfunction as a result of transfusion-induced iron-overload and oxidative stress associated with the disease. Taking the current gaps in knowledge pertaining to MDS-related fatigue into account, the objective of this study is to improve understanding on the aetiology fatigue in MDS patients. To achieve this aim, the study will measure a comprehensive group of patient-reported and disease-related outcomes: i) prior to blood transfusion therapy when Hb levels are low and; ii) following blood transfusion therapy, when Hb levels have been increased. Results from the post-transfusion tests will be analyzed to determine which participants remain fatigued despite an increase in Hb, and which participants shown an improvement in fatigue.

ELIGIBILITY:
Inclusion Criteria:

* Patient affiliated to a social security regimen or beneficiary of the same
* Signed written informed consent form
* Patient, ≥ 18 years-old, with established diagnosis of myelodysplastic syndrome with low or intermediate-1 risk cytogenetic profile
* FACIT-F score ≤ 34,
* Indication of blood transfusion.

Exclusion Criteria:

* Contra-indication to experimental procedures and/or physical exercise,
* Concomitant cancer diagnosis,
* Patient under guardianship or deprived of his liberty or any condition that may affect the patient's ability to understand and sign the informed consent
* Refusing participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2020-10-20 (Actual); Primary Completion 2020-10-20 (Actual); Study Completion 2020-10-20 (Actual)

PRIMARY OUTCOMES:
Measurement of Fatigue using FACIT-F questionnaire | 10 days
  Measurement of Fatigue will be performed using FACIT-F questionnaire. This is a questionnaire with 13 questions about which the patient is positioned on a Likert scale ranging from 1 to 5 (1 = quite, 5 = not at all). By adding the answers, a score out of 65 is obtained. Unlike other scales the higher the score the less the patient is tired. As an indication, the non-sick average positions is 40.1 on this scale.

CONTACTS AND LOCATIONS:
Overall Officials: Denis Guyotat, PhD, Principal Investigator — CHU de Saint-Etienne
Locations (1):
- CHU de Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No